CLINICAL TRIAL: NCT06761716
Title: Neuropsychophysiological Comparison of Ericksonian Hypnotherapy and Cognitive Behavioral Therapy in Patients Diagnosed With Post-Traumatic Stress Disorder: A Protocol and Pilot Study of Two Armed Open Label Randomized Clinical Trial
Brief Title: Comparison of Ericksonian Hypnotherapy and CBT in PTSD: A Clinical Trial
Acronym: NEPTUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Selami Varol Ülker, Director, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61351342/020-395
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: PTSD
Keywords: Post-traumatic stress disorder (PTSD); Ericksonian Hypnotherapy; Cognitive Behavioral Therapy (CBT); Neuropsychophysiology; EEG (Electroencephalography); GSR (Galvanic Skin Response); Heart Rate (HR); Trauma Therapy; Randomized Clinical Trial (RCT); Psychological Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with three groups:
  Ericksonian Hypnotherapy (EH) Group: 12 weekly 50-minute sessions focusing on hypnotic suggestions for PTSD symptom relief.
  Cognitive Behavioral Therapy (CBT) Group: 12 weekly 50-minute sessions using cognitive and behavioral techniques for PTSD management.
  Control Group: No therapeutic intervention; participants undergo baseline and post-study assessments only.
  Primary Outcome: Reduction in PTSD symptom severity (PCL-5, BDI-II, BAI). Secondary Outcome: Changes in neurophysiological and physiological markers (EEG, GSR, HR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ericksonian Hypnotherapy (EH) Arm (Experimental): Participants will receive 12 weekly sessions of 50 minutes each, focusing on tailored hypnotic suggestions and subconscious communication techniques specifically designed to address PTSD symptoms.
  Interventions: Behavioral: Ericksonian Hypnotherapy
- Cognitive Behavioral Therapy (CBT) Arm (Active Comparator): Participants will receive 12 weekly sessions of 50 minutes each, utilizing cognitive restructuring, exposure exercises, and behavioral interventions to reduce PTSD symptoms.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Control Group (No Intervention): Participants in the control group will not receive any therapeutic intervention. They will undergo baseline and post-study assessments using neuropsychophysiological measures (EEG, GSR, HR) and psychological scales (PCL-5, BDI-II, BAI) to monitor changes over time without active treatment.

INTERVENTIONS:
Behavioral: Ericksonian Hypnotherapy — Participants in this group will receive 12 weekly sessions of 50 minutes each. The therapy will focus on tailored hypnotic suggestions, subconscious communication techniques, and trauma-focused interventions specifically designed to address PTSD symptoms. Sessions will be conducted by a certified hypnotherapist under clinical supervision.
  Arms: Ericksonian Hypnotherapy (EH) Arm
Behavioral: Cognitive Behavioral Therapy — Participants in this group will receive 12 weekly sessions of 50 minutes each. The therapy will utilize cognitive restructuring techniques, exposure exercises, and behavioral interventions aimed at reducing PTSD symptoms. Sessions will be led by a licensed psychotherapist trained in trauma-focused CBT.
  Arms: Cognitive Behavioral Therapy (CBT) Arm

SUMMARY:
Brief Summary (Plain Language) The goal of this clinical trial is to compare the effects of Ericksonian Hypnotherapy and Cognitive Behavioral Therapy (CBT) on people diagnosed with Post-Traumatic Stress Disorder (PTSD). The study will also evaluate how these therapies impact brain activity, skin conductance, and heart rate.

The main questions it aims to answer are:

Does Ericksonian Hypnotherapy reduce PTSD symptoms as effectively as CBT? Do these therapies affect brain activity, skin conductance, and heart rate differently?

Participants will be randomly assigned to one of two therapy groups:

Ericksonian Hypnotherapy Group: Weekly 50-minute sessions for 12 weeks. CBT Group: Weekly 50-minute sessions for 12 weeks. To assess physiological and emotional responses, researchers will measure brain activity (EEG), skin conductance (GSR), and heart rate (HR) at various points. These assessments include a guided discussion task where participants reflect on their trauma in a controlled therapeutic environment. This task allows researchers to evaluate emotional regulation and stress markers in real time.

This study aims to provide insight into the physiological and psychological impacts of both therapies on PTSD treatment, offering a deeper understanding of how these interventions influence neurophysiological stress responses.

DETAILED DESCRIPTION:
Study Description This clinical trial aims to compare the neuropsychophysiological effects of Ericksonian Hypnotherapy (EH) and Cognitive Behavioral Therapy (CBT) in individuals diagnosed with Post-Traumatic Stress Disorder (PTSD). Additionally, a control group will be included to observe natural changes without therapeutic intervention.

PTSD is a debilitating psychological condition triggered by exposure to traumatic events, characterized by symptoms such as intrusive thoughts, hyperarousal, avoidance behaviors, and negative mood states. Both CBT and EH have shown promise in alleviating PTSD symptoms, yet their comparative neuropsychophysiological impacts remain underexplored.

Study Design Participants: Individuals aged 18-60 diagnosed with PTSD.

Randomization: Participants will be randomly assigned to one of three groups:

Ericksonian Hypnotherapy Group (EH): 12 weekly sessions of 50 minutes each, focusing on subconscious communication, personalized hypnotic suggestions, and trauma symptom alleviation.

Cognitive Behavioral Therapy Group (CBT): 12 weekly sessions of 50 minutes each, utilizing structured cognitive restructuring, exposure exercises, and behavioral interventions.

Control Group: No therapeutic intervention will be provided. Participants will attend scheduled monitoring sessions for baseline and post-study assessments.

Assessment and Measurements

Neuropsychophysiological parameters will be assessed at two time points: pre-intervention (baseline) and post-intervention (after 12 weeks). Measurements will include:

Electroencephalography (EEG): To monitor brain activity patterns, focusing on prefrontal cortex activation and emotional regulation networks.

Galvanic Skin Response (GSR): To measure changes in autonomic nervous system activity and emotional arousal.

Heart Rate (HR): To evaluate cardiovascular responses and physiological stress markers.

Participants will also engage in a guided trauma discussion task during these assessments, where they reflect on their traumatic experiences in a controlled therapeutic environment. This task enhances the ecological validity of the neurophysiological data by eliciting real-time emotional and cognitive responses to trauma-related stimuli.

Psychological Scales: PTSD Checklist for DSM-5 (PCL-5), Beck Depression Inventory-II (BDI-II), and Beck Anxiety Inventory (BAI) will be used to assess symptom severity.

Study Objectives Primary Objective: Compare the effectiveness of EH and CBT in reducing PTSD symptom severity.

Secondary Objective: Evaluate differences in neuropsychophysiological responses (EEG, GSR, HR) between EH, CBT, and the control group.

Exploratory Objective: Determine if EH offers comparable or superior benefits to CBT in modulating neurophysiological and physiological stress markers.

Expected Outcomes Symptom Reduction: EH and CBT are hypothesized to significantly reduce PTSD symptoms compared to the control group.

Neurophysiological Differentiation: Differences in neurophysiological and physiological markers are expected between EH and CBT groups.

Minimal Control Improvement: The control group is expected to show minimal or no significant improvement in symptoms or physiological parameters.

This study aims to provide robust comparative data on the efficacy and neuropsychophysiological effects of EH and CBT in PTSD treatment, offering clinicians valuable insights into therapeutic decision-making. The findings will contribute to refining treatment protocols and advancing evidence-based mental health interventions.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-60 years. Diagnosed with Post-Traumatic Stress Disorder (PTSD) based on DSM-5 criteria. No current psychiatric medication usage. Not undergoing any other psychotherapeutic intervention during the study period.

Ability to attend all therapy sessions and assessments. Ability to provide written informed consent. No neurological disorders or cognitive impairments that could affect participation.

Exclusion Criteria:

Individuals under 18 or over 60 years of age. Current or past diagnosis of schizophrenia, bipolar disorder, or other severe psychiatric disorders.

Acute risk of harm from engaging in trauma discussions. Use of psychiatric medication within the last 3 months. Ongoing participation in other psychotherapeutic interventions. History of substance abuse or dependence in the past 12 months. Known neurological disorders (e.g., epilepsy, traumatic brain injury). Inability to provide informed consent or comply with study procedures. Pregnancy or breastfeeding. Severe cardiovascular conditions that might interfere with physiological assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Reduction in PTSD Symptom Severity | Baseline and Week 12
  Change in PTSD symptom severity, measured by the PTSD Checklist for DSM-5 (PCL-5). Scores will assess the frequency and intensity of PTSD symptoms.

SECONDARY OUTCOMES:
Changes in Brain Activity (EEG) | Baseline and Week 12
  Differences in prefrontal cortex activity, as assessed by electroencephalography (EEG), measured during baseline and Week 12 sessions. EEG metrics, including power in alpha and theta bands and activation in emotional regulation networks, will also be recorded during a guided trauma discussion task designed to elicit real-time emotional and cognitive responses to trauma-related stimuli.
Changes in Heart Rate (HR) | Baseline and Week 12
  Evaluation of heart rate (HR) changes as a physiological marker of stress. Measurements will include baseline and Week 12 resting HR, as well as HR fluctuations during a guided trauma discussion task to capture autonomic nervous system activity in response to real-time trauma-related emotional processing.
Reduction in Anxiety Symptoms | Baseline and Week 12
  Change in anxiety severity, assessed using the Beck Anxiety Inventory (BAI). Scores will reflect self-reported anxiety symptoms.
Reduction in Depression Symptoms | Baseline and Week 12
  Change in depression severity, assessed using the Beck Depression Inventory-II (BDI-II). Scores will evaluate the frequency and impact of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Selami Varol Ülker, Phd, Principal Investigator — Üsküdar University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University; Eda Yılmazer, Phd, Principal Investigator — Beykoz University; Gökben Hızlı Sayar, Prof, Study Chair — Üsküdar University
Locations (1):
- Üsküdar University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study will be shared, after de-identification, to ensure participant confidentiality. This includes neuropsychophysiological data (EEG, GSR, HR), psychological assessment scores (PCL-5, BDI-II, BAI), and sociodemographic information relevant to the study's objectives.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available after publication of the primary results in an SSCI-indexed journal and will remain accessible for 5 years.
Access Criteria: Data will be made available to qualified researchers upon submission of a methodologically sound proposal and approval by the principal investigator.